CLINICAL TRIAL: NCT01541540
Title: Reducing Risk With E-based Support for Adherence to Lifestyle Change in Hypertension
Brief Title: e-Counseling Promotes Blood Pressure Reduction and Therapeutic Lifestyle Change in Hypertension
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 11-0580-BE; NCT01792076 (obsolete NCT alias)
Record Dates: First submitted 2012-02-17; First posted 2012-03-01 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Distance Counseling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- e-Counseling plus Usual Care (Experimental)
  Interventions: Behavioral: e-Counseling plus Usual Care
- e-Info Control plus Usual Care (Active Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: e-Counseling plus Usual Care — 28 emails will be sent proactively over a 12-month period. Emails will be sent weekly for the first 4 months, biweekly from months 5 to 8, and monthly from months 9 to 12. Each email will contain an e-link to lifestyle counseling activities designed to enhance motivation and skill to initiate and maintain lifestyle change. e-Counseling includes video-based education and counseling as well as e-tools to self-monitor and reinforce adherence to self-management behavior for exercise, diet, prescribed medications and smoke-free living.
  Arms: e-Counseling plus Usual Care
Behavioral: Control — The control group will receive general educational material on heart healthy living. 28 emails will be sent proactively over a 12-month period. Emails will be sent weekly for the first 4 months, biweekly from months 5 to 8, and monthly from months 9 to 12.
  Arms: e-Info Control plus Usual Care

SUMMARY:
This proposed clinical trial, REACH, will enroll 538 persons with hypertension. All subjects will continue with their prescribed medications. Our main objective is to assess whether preventive e-counseling (provided through a website of the Heart and Stroke Foundation) improves blood pressure and cardiovascular risk status over a 12-month interval. REACH will also evaluate improvement in lifestyle behaviors that include diet, exercise, smoking, and adherence to prescribed medications. Finally, we will quantify the amount of e-counseling support that is required during REACH to evoke a significant reduction in blood pressure. It is hypothesized that e-Counseling (vs. Control) will significantly improve blood pressure and lifestyle behaviours at the 12-month assessment. The findings of this trial will provide information that is critical to our understanding of how internet-based programs can help to improve blood pressure and to reduce the risk for cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Age: 35-74 years
* Diagnosis of hypertension: Medication or physician confirmation
* Baseline BP in lab: >=140/90 (if no meds); >=130/85 (if on meds)
* If medications, prescription unchanged >=2 months Comprehension of English (oral and written)

Exclusion Criteria:

* diagnosis of clinically significant arrhythmia, sleep apnea, kidney disease, major psychiatric illness (eg. psychosis), alcohol or drug dependence in the previous year; institutional residence, or an inability to comprehend English

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2012-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 12-month
  Systolic blood pressure, diastolic blood pressure, pulse pressure
lipoprotein cholesterol | 12-month
  total, low-density, and total/high-density ratio
10-year absolute risk for Cardiovascular Heart Disease. | 12-month

SECONDARY OUTCOMES:
4-day step count recorded by accelerometry | 12-month
24-hour urinary sodium excretion | 12-month
salivary cotinine | 12-month
  smoke-free living measured by salivary cotinine. Measured only in smokers
Fruit and vegetable intake | 12-month
  Diet History Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Nolan, Ph.D, Principal Investigator — Behavioural Cardiology Research Unit, University Health Network
Locations (4):
- Canada (4):
  - Vancouver Coastal Health, Vancouver, British Columbia
  - London Health Science Center, London, Ontario
  - Grey Bruce Health Unit, Owen Sound, Ontario
  - University Health Network (Toronto Gen Hosp Site), Toronto, Ontario

REFERENCES:
- [Derived] Liu S, Tanaka R, Barr S, Nolan RP. Effects of self-guided e-counseling on health behaviors and blood pressure: Results of a randomized trial. Patient Educ Couns. 2020 Mar;103(3):635-641. doi: 10.1016/j.pec.2019.10.007. Epub 2019 Oct 19. PMID 31669047
- [Derived] Nolan RP, Feldman R, Dawes M, Kaczorowski J, Lynn H, Barr SI, MacPhail C, Thomas S, Goodman J, Eysenbach G, Liu S, Tanaka R, Surikova J. Randomized Controlled Trial of E-Counseling for Hypertension: REACH. Circ Cardiovasc Qual Outcomes. 2018 Jul;11(7):e004420. doi: 10.1161/CIRCOUTCOMES.117.004420. PMID 30006474
- [Derived] Tanaka R, Nolan RP. Psychobehavioral Profiles to Assist Tailoring of Interventions for Patients With Hypertension: Latent Profile Analysis. J Med Internet Res. 2018 May 11;20(5):e149. doi: 10.2196/jmir.8757. PMID 29752248
- [Derived] Nolan RP, Liu S, Feldman R, Dawes M, Barr S, Lynn H, Gwardy-Sridhar F, Thomas SG, Goodman J, Oh P, Kaczorowski J, Chessex C, Hachinski V, Shoemaker K. Reducing risk with e-based support for adherence to lifestyle change in hypertension (REACH): protocol for a multicentred randomised controlled trial. BMJ Open. 2013 Aug 21;3(8):e003547. doi: 10.1136/bmjopen-2013-003547. PMID 23965936